CLINICAL TRIAL: NCT05189561
Title: Near-infrared Spectroscopy (NIRS) for Intracranial Hematoma Detection in Traumatic Head Injury
Brief Title: Near-infrared Spectroscopy (NIRS) for Intracranial Hematoma Detection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Mental Health and Neuro Sciences, India (Other)
Responsible Party: Principal Investigator, Dhaval Shukla, Prof. of Neurosurgery, National Institute of Mental Health and Neuro Sciences, India
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: NIMHANS/24thIEC(BS&NSDIV)
Record Dates: First submitted 2021-11-26; First posted 2022-01-12 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-02

CONDITIONS: Traumatic Brain Injury
Keywords: traumatic brain injury; traumatic intracranial hematoma; extradural hematoma; subdural hematoma; cerebral contusion; near-infrared spectroscopy
MeSH Terms: conditions — Brain Injuries, Traumatic; Intracranial Hemorrhage, Traumatic; Hematoma, Epidural, Spinal; Hematoma, Subdural; Brain Contusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cerebo® (Experimental): Participants undergoing scanning using NIRS device.
  Interventions: Other: near-infrared scanner

INTERVENTIONS:
Other: near-infrared scanner — Tests to be administered: Near Infra-Red Scanning of the head at the bedside.
  Time taken for testing: Two minutes
  Biological samples collected: None
  Frequency of testing/collection: Once
  Risks for the participants while being tested: None
  Other Names: Cerebo

SUMMARY:
Traumatic brain injury is a common neurosurgical emergency managed in all tertiary and secondary hospitals. Detecting the underlying pathology is a major challenge especially for surgical cases. The outcome differs if the early intervention is performed. Near-infrared spectroscopy (NIRS) based device will detect the hematoma at the bedside. It is not the replacement of a CT scan but can help in triage. This is a large-scale prospective study to establish the role of NIRS device in detecting intracerebral hematoma and correlate the finding with CT scan finding.

DETAILED DESCRIPTION:
The light used in the near-infrared spectrum, especially between 700 and 1000 nm, is able to penetrate the human tissue 'optical window'. Once the light has penetrated into the tissue, it is either scattered or absorbed. Light is mostly scattered by bones, skin and cerebral white matter. However, red blood cells, which represent roughly have a low scattering effect and high absorption. Utilising this principle, the emitter and detector could be used to measure the light scattered by the tissues. The 'optical density' of the tissue is calculated and by comparing the left and right hemispheres in the eight contralateral locations of the brain lobes where lesions with extravascular accumulation of haemoglobin can be detected. A NIRS device named Cerebo® was developed by Bioscan Research, Ahmedabad, India. It is a low power non risky device that can screen the patient's head multiple times without causing any side effect. The built in safety features in Cerebo® make it fail safe system for intentional as well as accidental exposure to laser beam. The average power and total power dissipation is very low. The system poses no risk to the patients who will be included in the study.

So far the overall results of detection rate of hematoma using NIRS device are contradictory. It is not the replacement of a CT scan but can help in triage. In the present research the investigators plan to do a large scale prospective study to establish the role of NIRS device in detecting intracerebral hematoma and correlate the finding with CT scan findings.

ELIGIBILITY:
Inclusion Criteria:

* Acute traumatic brain injury patients reaching the hospital

Exclusion Criteria:

* Major scalp laceration or active bleeding.
* Significant extracranial hematoma.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2021-08-24 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
Detection rate of intracranial hematoma | Immediately after the test
  To evaluate detection rate of intracranial hematoma using NIRS device Cerebo®, (Bioscan Research, Ahmedabad, India) in hospital.

SECONDARY OUTCOMES:
Detection rate of clinically significant intracranial hematoma | Immediately after the test
  To evaluate detection rate of clinically significant intracranial hematoma using NIRS device Cerebo®, (Bioscan Research, Ahmedabad, India), which requires admission or surgical intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Dhaval Shukla, MCh, Principal Investigator — National Institute of Mental Health and Neuro Sciences, India
Locations (1):
- NIMHANS, Bangalore, Karnataka, India

DOCUMENTS (1):
  • Study Protocol (2020-09-19): https://cdn.clinicaltrials.gov/large-docs/61/NCT05189561/Prot_000.pdf